CLINICAL TRIAL: NCT00121199
Title: Phase II Trial of Standard Dose Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (CHOP) and Rituximab Plus Bevacizumab for Advanced Stage Diffuse Large B-Cell NHL
Brief Title: Combination Chemo, Rituximab, and Bevacizumab in Older Patients With Stage II-IV Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03062; NCI-2012-03062 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S0515 (Other: SWOG); S0515 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2012-12

CONDITIONS: Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Bevacizumab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

ARMS (1):
- Treatment (CHOP, rituximab, bevacizumab) (Experimental): Patients receive rituximab IV, bevacizumab IV over 30-90 minutes, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1. Patients also receive oral prednisone on days 1-5. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Biological: bevacizumab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving combination chemotherapy together with rituximab and bevacizumab works in treating older patients with stage II, stage III, or stage IV diffuse large B-cell lymphoma. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Monoclonal antibodies, such as rituximab and bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bevacizumab may also stop the growth of cancer cells by blocking blood flow to the cancer. Giving combination chemotherapy together with monoclonal antibodies may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the 1-year progression-free survival rate in patients with advanced stage diffuse large B-cell NHL treated with CHOP - rituximab - bevacizumab.

II. To estimate the response rate (complete, complete unconfirmed, and partial) and 2-year progression-free survival of this regimen in patients with advanced stage diffuse large B-cell NHL.

III. To evaluate the toxicities associated with this regimen. IV. To correlate angiogenic biomarkers with patient outcome.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV, bevacizumab IV over 30-90 minutes, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1. Patients also receive oral prednisone on days 1-5. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at least every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have previously untreated Stage III, IV, or bulky Stage II diffuse large B-cell non-Hodgkin's lymphoma which is positive for CD20; a report providing confirmation of CD20 expression must be submitted
* Pathology Review: Adequate sections from the original diagnostic specimen must be available for submission for review by the SWOG Lymphoma Pathology Laboratory; an adequate biopsy requires sufficient tissue to establish the architecture and a REAL or WHO histologic subtype with certainty; thus, core biopsies, especially multiple core biopsies may be adequate; whereas, needle aspirations or cytologies are not adequate
* Specimens for analysis of angiogenic markers must be submitted to the University of Arizona
* All patients must have bidimensionally measurable disease documented within 28 days prior to registration; patients with non-measurable disease in addition to measurable disease must have all nonmeasurable disease assessed within 42 days prior to registration
* Patients must have a unilateral or bilateral bone marrow aspirate and biopsy performed within 42 days prior to registration
* Patients must have a CT scan of the chest/abdomen and pelvis performed within 28 days prior to registration
* Patients must not have clinical evidence of central nervous system involvement by lymphoma; any laboratory or radiographic tests performed to assess CNS involvement must be negative within 42 days of registration
* Patients may not have a previous diagnosis of indolent lymphoma (histologic transformation or mixed histologies with an indolent or nodular component are ineligible)
* Patients must not have received prior chemotherapy, radiation, or antibody-based therapy for lymphoma
* Patients must have a Zubrod performance status of 0 - 2
* Serum LDH must be measured within 28 days prior to registration
* Patients must have a cardiac ejection fraction >= 45% by MUGA scan or a 2-d ECHO with no significant abnormalities within 42 days prior to registration
* Absolute neutrophil count > 1,000/mcL obtained within 28 days prior to registration
* Platelet count > 100,000/mcL obtained within 28 days prior to registration
* Serum creatinine < 2 x the institutional upper limit of normal within 28 days prior to registration
* Patients must have urine proteinuria screened by dipstick or urine analysis within 28 days prior to registration; in patients with proteinuria >= +1 or urine protein:creatinine ratio >= 1.0, a 24 hour urine protein should be obtained and the level < 1gm/24 hours to be eligible
* Patients must not have a history of hypersensitivity reaction to products containing Polysorbate 20 (Tween 20), Chinese hamster ovary cell products, or recombinant human antibodies
* Patients known to be HIV-positive, or who have a history of solid organ transplantation are ineligible due to the concern over immunosuppression associated with B-cell depletion; patients at high risk of Hepatitis B virus infection should be screened before initiation of rituximab
* Patients must not have uncontrolled hypertension
* Patients with a history of prior myocardial infarction, unstable angina, stroke, or arterial thrombosis within 6 months are ineligible
* Patients with clinically significant peripheral vascular disease, a serious or non-healing wound, ulcer, or bone fracture, or a bleeding diathesis/coagulopathy are ineligible
* Patients with a history of venous thrombosis requiring full-dose anticoagulation or currently receiving anticoagulation therapy may be eligible provided that the following criteria are met:

  * The patient must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on a stable dose of LMW heparin
  * The patient must not have bleeding or pathological conditions that carry a high risk of bleeding (e.g. tumor involving major vessels, known varices)
* Patients who have had a major surgical procedure or traumatic injury within 28 days prior to registration or anticipation of major surgical procedure during the course of therapy are ineligible
* Patients with a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months are ineligible
* Patients requiring continuous supplemental oxygen therapy are ineligible
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer for which the patient has been disease-free for five years
* Pregnant or nursing women may not participate in this study due to the potential for congenital abnormalities, and of harm to nursing infants due to this treatment regimen; women or men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during the study period and for at least 6 months after the completion of therapy
* If Day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Stopeck, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- SWOG, Portland, Oregon, United States

REFERENCES:
- [Derived] Stopeck AT, Unger JM, Rimsza LM, LeBlanc M, Farnsworth B, Iannone M, Glenn MJ, Fisher RI, Miller TP. A phase 2 trial of standard-dose cyclophosphamide, doxorubicin, vincristine, prednisone (CHOP) and rituximab plus bevacizumab for patients with newly diagnosed diffuse large B-cell non-Hodgkin lymphoma: SWOG 0515. Blood. 2012 Aug 9;120(6):1210-7. doi: 10.1182/blood-2012-04-423079. Epub 2012 Jun 25. PMID 22734071

RESULTS

PARTICIPANT FLOW:
Groups:
- CHOP + Rituximab + Bevacizumab: Treatment with CHOP, rituximab, and bevacizumab will be administered every 21 days for a maximum of 8 cycles (one cycle is defined as a single 21 day course of treatment). Bevacizumab and rituximab will be given before chemotherapy.
Period: Overall Study
Arm/Group | CHOP + Rituximab + Bevacizumab
Started | 73
Eligible | 64
Eligible and Began Protocol Therapy | 64
Completed | 45
Not Completed | 28
Not completed — Adverse Event | 11
Not completed — Refusal Unrelated to Adverse Event | 1
Not completed — Progression/Relapse | 1
Not completed — Death | 3
Not completed — Other - Not Protocol Specified | 3
Not completed — Ineligible | 9

BASELINE CHARACTERISTICS:
Arm/Group | CHOP + Rituximab + Bevacizumab
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 67.6 [21.8 to 84.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Secondary Outcome: Objective Response (Confirmed and Unconfirmed Complete Response (CR) or Partial Response (PR))
Description: Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow(BM) must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRU) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM. Partial Response(PR) is a 50% decrease in the SPD for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: After Cycle 4 (Day 64) but prior to Cycle 5 (Day 85) and after Cycle 8 (Day 181). After completion of protocol treatment, every 6 months for 2 years, then annually for a maximum of five years.
Population: All patients who started treatment were included in the analysis
Measure: Number; unit: participants
Arm/Group | CHOP + Rituximab + Bevacizumab
Number analyzed (Participants) | 64
participants
  Complete Response (CR) | 22
  Partial Response (PR) | 20
  Unconfirmed Complete Response (UCR) | 6
  Unconfirmed Partial Response (UPR) | 1
  No Response | 15

2. Primary Outcome: Progression-free Survival at 1 Year
Description: Measured from time of registration to date of of first observation of progression/relapse, or death due to any cause, or last contact date
Time Frame: 0-1 year
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHOP + Rituximab + Bevacizumab
Number analyzed (Participants) | 64
percentage of participants | 77 [66 to 87]

3. Primary Outcome: Progression-free Survival at 2 Year
Description: as for outcome 2
Time Frame: 0-2 years
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHOP + Rituximab + Bevacizumab
Number analyzed (Participants) | 64
percentage of participants | 69 [57 to 80]

4. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Patients were assessed for adverse events after every cycle (1 cycle = 21 days) of protocol treatment
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | CHOP + Rituximab + Bevacizumab
Number analyzed (Participants) | 63
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1
  Allergic reaction/hypersensitivity | 1
  Anorexia | 5
  Cardiac General-Other (Specify) | 1
  Cardiac troponin I (cTnI) | 1
  Cardiopulmonary arrest, cause unknown (non-fatal) | 1
  Constipation | 2
  Dehydration | 1
  Distention/bloating, abdominal | 1
  Dry mouth/salivary gland (xerostomia) | 1
  Dyspnea (shortness of breath) | 3
  Fatigue (asthenia, lethargy, malaise) | 8
  Febrile neutropenia | 11
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 1
  Glucose, serum-high (hyperglycemia) | 2
  Hemoglobin | 8
  Hemolysis | 1
  Hemorrhage, GI - Colon | 1
  Hemorrhage, pulmonary/upper respiratory - Nose | 2
  Hypertension | 4
  Hypotension | 2
  Hypoxia | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Ab NOS | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 1
  Insomnia | 1
  Left ventricular diastolic dysfunction | 1
  Left ventricular systolic dysfunction | 3
  Leukocytes (total WBC) | 28
  Lymphopenia | 10
  Mucositis/stomatitis (clinical exam) - Oral cavity | 2
  Muscle weakness, not d/t neuropathy - body/general | 2
  Nausea | 2
  Neuropathy: motor | 3
  Neuropathy: sensory | 1
  Neutrophils/granulocytes (ANC/AGC) | 33
  Obstruction, GI - Jejunum | 1
  Pain - Abdomen NOS | 4
  Pain - Bone | 1
  Pain - Throat/pharynx/larynx | 1
  Perforation, GI - Jejunum | 2
  Perforation, GI - Small bowel NOS | 1
  Perforation, GI - Stomach | 1
  Platelets | 12
  Pneumonitis/pulmonary infiltrates | 1
  Pneumothorax | 1
  Potassium, serum-low (hypokalemia) | 2
  Pruritus/itching | 1
  Pulmonary/Upper Respiratory-Other (Specify) | 2
  Renal failure | 1
  Sodium, serum-low (hyponatremia) | 3
  Somnolence/depressed level of consciousness | 1
  Sudden death | 2
  Thrombosis/thrombus/embolism | 4
  Voice changes/dysarthria | 1
  Vomiting | 1
  Weight loss | 1

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events after every cycle (1 cycle = 21 days) of protocol treatment
Arm/Group | CHOP + Rituximab + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 27/63
Other Adverse Events (participants affected / at risk) | 60/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CHOP + Rituximab + Bevacizumab (N=63)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Hemorrhage, GI - Colon (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) - Esophagus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Perforation, GI - Jejunum (Gastrointestinal disorders) | 2
Perforation, GI - Small bowel NOS (Gastrointestinal disorders) | 1
Perforation, GI - Stomach (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3
Pain-Other (Specify) (General disorders) | 1
Sudden death (General disorders) | 2
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Skin (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Lymphatic (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Perit cav (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Leukocytes (total WBC) (Investigations) | 4
Lymphopenia (Investigations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7
Platelets (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 1
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuropathy: motor (Nervous system disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CHOP + Rituximab + Bevacizumab (N=63)
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Hemoglobin (Blood and lymphatic system disorders) | 42
Left ventricular systolic dysfunction (Cardiac disorders) | 8
Constipation (Gastrointestinal disorders) | 30
Diarrhea (Gastrointestinal disorders) | 19
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 5
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 4
Heartburn/dyspepsia (Gastrointestinal disorders) | 7
Hemorrhoids (Gastrointestinal disorders) | 4
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 20
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 25
Pain - Abdomen NOS (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 10
Edema: limb (General disorders) | 9
Fatigue (asthenia, lethargy, malaise) (General disorders) | 47
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 13
Pain-Other (Specify) (General disorders) | 9
Rigors/chills (General disorders) | 12
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 4
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 13
AST, SGOT (Investigations) | 15
Alkaline phosphatase (Investigations) | 10
Bilirubin (hyperbilirubinemia) (Investigations) | 6
Creatinine (Investigations) | 8
Leukocytes (total WBC) (Investigations) | 32
Lymphopenia (Investigations) | 16
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 32
Platelets (Investigations) | 26
Weight loss (Investigations) | 14
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 18
Anorexia (Metabolism and nutrition disorders) | 24
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 14
Dehydration (Metabolism and nutrition disorders) | 8
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 27
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 9
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 17
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 5
Pain - Back (Musculoskeletal and connective tissue disorders) | 14
Pain - Bone (Musculoskeletal and connective tissue disorders) | 4
Pain - Joint (Musculoskeletal and connective tissue disorders) | 10
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 6
Neuropathy: motor (Nervous system disorders) | 5
Neuropathy: sensory (Nervous system disorders) | 32
Pain - Head/headache (Nervous system disorders) | 14
Taste alteration (dysgeusia) (Nervous system disorders) | 11
Insomnia (Psychiatric disorders) | 11
Mood alteration - anxiety (Psychiatric disorders) | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 19
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 15
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 5
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 6
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 4
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 25
Nail changes (Skin and subcutaneous tissue disorders) | 4
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less